CLINICAL TRIAL: NCT00988065
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Incidence of Hypersensitivity After Repeated Single Dose Administrations of Sugammadex (SCH 900616) in Healthy Subjects
Brief Title: Sugammadex Hypersensitivity Study (Study P06042)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06042; EUDRACT: 2009-012014-40
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugammadex 4 mg/kg (Experimental): Participants were to receive one dose of sugammadex 4 mg/kg intravenous bolus injection on Day 8, Day 36, and Day 78 of the study.
  Interventions: Drug: Placebo run-in dose; Drug: Sugammadex 4 mg/kg
- Sugammadex 16 mg/kg (Experimental): Participants were to receive one dose of sugammadex 16 mg/kg intravenous bolus injection on Day 8, Day 36, and Day 78 of the study.
  Interventions: Drug: Placebo run-in dose; Drug: Sugammadex 16 mg/kg
- Placebo (Placebo Comparator): Participants were to receive one dose of placebo intravenous bolus injection on Day 8, Day 36, and Day 78 of the study.
  Interventions: Drug: Placebo run-in dose; Drug: Placebo

INTERVENTIONS:
Drug: Placebo run-in dose — Single-blind placebo intravenous bolus injection on Day 1 of the study, 7 days prior to randomization
Drug: Sugammadex 4 mg/kg — Sugammadex 4 mg/kg intravenous bolus injection on Day 8, Day 36, and Day 78 of the study
  Other Names: SCH 900616, Org 25969, Bridion®
  Arms: Sugammadex 4 mg/kg
Drug: Sugammadex 16 mg/kg — Sugammadex 16 mg/kg intravenous bolus injection on Day 8, Day 36, and Day 78 of the study
  Other Names: SCH 900616, Org 25969, Bridion®
  Arms: Sugammadex 16 mg/kg
Drug: Placebo — Placebo intravenous bolus injection on Day 8, Day 36, and Day 78 of the study
  Arms: Placebo

SUMMARY:
This trial was conducted to study the potential for hypersensitivity symptoms at the time of initial exposure to sugammadex and upon repeat exposure, since it was unknown whether the frequency or severity of hypersensitivity symptoms may worsen at repeat exposure over a prolonged period.

In total 450 participants (all healthy subjects) were to be randomized to receive one of three study treatments: three repeated doses of either sugammadex 4 mg/kg, sugammadex 16 mg/kg, or placebo. Participants were to receive one dose of study treatment on Day 8, Day 36, and Day 78 of the study in order to determine the safety of each treatment dose.

DETAILED DESCRIPTION:
All subjects were to be admitted to the study center the day before each scheduled dose and were to leave the unit the morning of the day after each dose. In cases of suspected hypersensitivity symptoms, healthy subjects were to remain confined to the study center until all signs and symptoms regressed, the subject was stable, and the investigator considered it safe for the subject to leave the study center. Four sites participated in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Serum tryptase <=11.4 mcg/L and fasting triglyceride levels within normal limits
* Safety laboratory tests and vital signs must have been within normal limits
* Screening electrocardiogram must have been clinically acceptable and parameters within normal limits
* Body Mass Index between 19 and 32 kg/m^2
* Females must have agreed to use contraceptives
* Other certain administrative criteria as described in the protocol

Exclusion Criteria:

* Females who were pregnant or intending to become pregnant
* Subjects who would not be able to participate optimally in the study, in the opinion of the investigator
* Certain surgical or medical conditions, recent infections, or mental instability
* Positive test for certain drugs or history of alcohol or drug abuse
* Positive test for hepatitis B, hepatitis C, or Human Immunodeficiency Virus (HIV)
* Blood donation in the past 60 days
* A history of unexplained reaction or hypersensitivity reaction during previous surgery and/or anesthesia
* History of anaphylaxis from any cause, suspected history of hypersensitivity to cyclodextrins, or multiple drug hypersensitivities
* Heavy smoker
* Received certain medications in the past
* History of allergy, hypersensitivity, or intolerance to epinephrine at greater risk of developing adverse reactions after epinephrine administration
* Other certain administrative criteria as described in the protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 448 (Actual)
Dates: Start 2009-09-06 (Actual); Primary Completion 2010-04-13 (Actual); Study Completion 2010-04-13 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] de Kam PJ, Nolte H, Good S, Yunan M, Williams-Herman DE, Burggraaf J, Kluft C, Adkinson NF, Cullen C, Skov PS, Levy JH, van den Dobbelsteen DJ, van Heumen ELGM, van Meel FCM, Glassner D, Woo T, Min KC, Peeters PAM. Sugammadex hypersensitivity and underlying mechanisms: a randomised study of healthy non-anaesthetised volunteers. Br J Anaesth. 2018 Oct;121(4):758-767. doi: 10.1016/j.bja.2018.05.057. Epub 2018 Jul 13. PMID 30236238

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 480 participants received a single-blind placebo dose 7 days prior to randomization. Of these 480 participants, 448 were randomized to double-blind treatment.
Period: Overall Study
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Started | 148 (Randomized to double-blind treatment) | 150 (Randomized to double-blind treatment) | 150 (Randomized to double-blind treatment)
Received First Randomized Dose | 148 | 150 | 150
Received Second Randomized Dose | 139 | 135 | 145
Received Third Randomized Dose | 135 | 127 | 135
Completed | 135 | 127 | 135
Not Completed | 13 | 23 | 15
Not completed — Adverse Event | 4 | 10 | 2
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Subject withdrew consent | 3 | 5 | 2
Not completed — Noncompliance with protocol | 5 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo | Total
Number analyzed (Participants) | 148 | 150 | 150 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (10.6) | 33.2 (10.2) | 33.8 (10.8) | 33.8 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 73 | 75 | 218
  Male | 78 | 77 | 75 | 230

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Adjudicated Hypersensitivity Signs/Symptoms, for Each Sugammadex Dose Group and Placebo.
Description: Hypersensitivity signs/symptoms were systematically collected for each subject by the investigator. Suspected cases of hypersensitivity signs/symptoms were sent to the independent Adjudication Committee (comprised of anesthesiologists & allergists/immunologists) for blinded review and determination of adjudicated hypersensitivity &/or anaphylaxis based on expert evaluation of all clinical data from the healthy subject.
  The percentages of subjects who had adjudicated hypersensitivity at any dose (dose 1/Day 8, dose 2/Day 36, or dose 3/Day 78) were compared between the 3 treatment groups.
Time Frame: Day 8, Day 36, and Day 78 of the study
Population: All-Subjects as treated (i.e., who received at least one dose of randomized study medication).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Number analyzed (Participants) | 148 | 150 | 150
percentage of participants | 0.7 [0.0 to 3.7] | 4.7 [1.9 to 9.4] | 0 [0 to 2.4]
Statistical Analysis 1: Comparison: Sugammadex 4 mg/kg vs Placebo; Test type: Superiority or Other; Difference in event rates = 0.7, 95% CI [-1.8 to 3.7] — 95% confidence interval for the difference in event rates (treatment group minus placebo) according to Miettinen and Nurminen (Statistics in Medicine 1985; 4:213-226)
Statistical Analysis 2: Comparison: Sugammadex 16 mg/kg vs Placebo; Test type: Superiority or Other; Difference in event rates = 4.7, 95% CI [2.1 to 9.3] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: The Percentage of Participants With Adjudicated Anaphylaxis According to the Definition by Sampson et al., for Each Sugammadex Dose Group and Placebo.
Description: The Adjudication Committee evaluated each case to determine whether the subject's hypersensitivity sign/symptoms fulfilled the definition of anaphylaxis according to the criteria defined by the Symposium on the Definition and Management of Anaphylaxis as described by Sampson et al. (J Allergy Clin Immunol 2006; 117:391-7).
  The percentages of subjects who had adjudicated anaphylaxis according to the Sampson Criteria at any dose (dose 1 [~Day 8], dose 2 [~Day 36], or dose 3 [Day ~78]) were compared between the 3 treatment groups.
Time Frame: Day 8, Day 36, and Day 78 of the study
Population: All-Subjects as treated (i.e., who received at least one dose of randomized study medication).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Number analyzed (Participants) | 148 | 150 | 150
percentage of participants | 0 [0 to 2.5] | 0.7 [0.0 to 3.7] | 0 [0 to 2.4]
Statistical Analysis 1: Comparison: Sugammadex 16 mg/kg vs Placebo; Test type: Superiority or Other; Difference in event rates = 0.7, 95% CI [-1.8 to 3.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Placebo; Test type: Superiority or Other; Difference in event rates = 0, 95% CI [-2.5 to 2.5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: The Percentage of Participants With Each of the 3 Levels of Diagnostic Certainty of Adjudicated Anaphylaxis According to the Definition by Rüggeberg et al., for Each Sugammadex Dose Group and Placebo.
Description: The Adjudication Committee evaluated each case to determine anaphylaxis according to the criteria put forth by the guidelines of the Brighton Collaboration Anaphylaxis Working Group as described by Rüggeberg et al. (Vaccine 2007; 25:5675-5684).
  Level 1 represents the highest level of certainty of anaphylaxis and level 3 the lowest level of certainty.
  The percentages of subjects who had adjudicated anaphylaxis according to the Rüggeberg Criteria at any dose (dose 1 [~Day 8], dose 2 [~Day 36], or dose 3 [Day ~78]) were compared between the 3 treatment groups.
Time Frame: Day 8, Day 36, and Day 78 of the study
Population: All-Subjects as treated (i.e., who received at least one dose of randomized study medication).
Measure: Number; unit: percentage of participants
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Number analyzed (Participants) | 148 | 150 | 150
percentage of participants
  Level 1 | 0 | 0.7 | 0
  Level 2 | 0 | 1.3 | 0
  Level 3 | 0 | 0 | 0
  Level 1 or Level 2 | 0 | 2.0 | 0
Statistical Analysis 1: Comparison: Sugammadex 16 mg/kg vs Placebo; Comparison of participants who had Level 1 or Level 2 diagnostic certainty; Test type: Superiority or Other; Difference in event rates = 2.0, 95% CI [-0.5 to 5.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sugammadex 4 mg/kg vs Placebo; Comparison of participants who had Level 1 or Level 2 diagnostic certainty; Test type: Superiority or Other; Difference in event rates = 0, 95% CI [-2.5 to 2.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: The Percentage of Participants With Adjudicated Hypersensitivity Signs/Symptoms After Each Randomized Dose of Study Treatment, for Each Sugammadex Dose Group and Placebo.
Description: Hypersensitivity signs/symptoms were systematically collected for each subject by the investigator. Suspected cases of hypersensitivity signs/symptoms were sent to the independent Adjudication Committee (comprised of anesthesiologists & allergists/immunologists) for blinded review & determination of adjudicated hypersensitivity &/or anaphylaxis based on expert evaluation of all clinical data from the healthy subject.
  The percentages of subjects who had adjudicated hypersensitivity (dose 1/Day 8, dose 2/Day 36, or dose 3/Day 78) are presented for each of the 3 treatment arms for each dose.
Time Frame: Day 8, Day 36, and Day 78 of the study
Population: All-Subjects as treated, per dose (i.e. who received the corresponding dose of randomized study medication).
Measure: Number; unit: percentage of participants
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Number analyzed (Participants) | 148 | 150 | 150
percentage of participants
  1st randomized dose | 0.7 | 4.0 | 0
  2nd randomized dose (n=139; n=135; n=145) | 0.7 | 1.5 | 0
  3rd randomized dose (n=135; n=127; n=135) | 0 | 0.8 | 0
  after any randomized dose | 0.7 | 4.7 | 0

5. Other Pre Specified Outcome: Percentage of Participants With an Adverse Event Suggestive of a Dose-dependent Trend That Also Exceeds a Frequency Threshold Above 5% in Any Treatment Arm (Including Both Serious and Non-serious Adverse Events).
Description: All adverse events from the study were reviewed for potential safety signals. The reported incidences suggestive of a dose-dependent trend and with a frequency threshold above 5% (including both serious and non-serious adverse events) are presented.
Time Frame: From first randomized dose (Day 8) up to 30 days after day of last randomized dose of study medication.
Population: All-Subjects as treated (i.e., who received at least one dose of randomized study medication).
Measure: Number; unit: percentage of participants
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Number analyzed (Participants) | 148 | 150 | 150
percentage of participants
  Flushing | 1.4 | 5.3 | 0.7
  Nausea | 5.4 | 16.0 | 1.3
  Dysgeusia | 3.4 | 21.3 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) that started after first dose of randomized study medication up to 30 days after day of last dose of randomized study medication, i.e. the "Treatment-emergent" AEs.
Arm/Group | Sugammadex 4 mg/kg | Sugammadex 16 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/148 | 2/150 | 1/150
Other Adverse Events (participants affected / at risk) | 35/148 | 64/150 | 33/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 4 mg/kg (N=148) | Sugammadex 16 mg/kg (N=150) | Placebo (N=150)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 4 mg/kg (N=148) | Sugammadex 16 mg/kg (N=150) | Placebo (N=150)
Nausea (Gastrointestinal disorders) | 8 (11) | 24 (34) | 2 (3)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10) | 13 (15)
Dysgeusia (Nervous system disorders) | 5 (8) | 32 (43) | 0 (0)
Headache (Nervous system disorders) | 17 (20) | 19 (23) | 16 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 9 (9)

LIMITATIONS AND CAVEATS:
Results from this study in healthy/conscious subjects may not be fully applicable to anesthetized patient settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may not publish/publicly present interim results without prior consent of Sponsor. Any materials that report results of the study must be sent to Sponsor 45 days prior to submission for publication/presentation. Sponsor has right to review and comment. In case of any disagreements concerning appropriateness of the materials, investigator and Sponsor must meet to make a good faith effort to discuss/resolve the issues or disagreement, prior to submission for publication/presentation.